CLINICAL TRIAL: NCT05679466
Title: An Investigator Initiated, Randomized, Double-blinded, Placebo-controlled Clinical Trial to Evaluate the Safety, Immunogenicity and Efficacy of the Recombinant Two-component COVID-19 Vaccine (CHO Cell) in Adults Aged 18 Years and Older
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yu Qin (Other)
Responsible Party: Sponsor-Investigator, Yu Qin, senior technologist, West China Second University Hospital
Organization: West China Second University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC611-IIT-1
Record Dates: First submitted 2023-01-09; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Prevention of COVID-19 Caused by SARS-CoV-2
MeSH Terms: interventions — Random Allocation; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReCOV (Active Comparator)
  Interventions: Biological: randomized, double-blinded, placebo-controlled
- ReCOV placebo (Placebo Comparator)
  Interventions: Biological: randomized, double-blinded, placebo-controlled

INTERVENTIONS:
Biological: randomized, double-blinded, placebo-controlled — Approximately 3300 participants will be enrolled, including an immunogenic subgroup of approximately 240. Approximately 10% to 15% of all subjects will be 60 years of age and older. Enrolled subjects will be stratified by age (18-59 years, 60 years and older), number of previous doses of COVID-19 vaccine (2 or 3 doses), and interval from the last previous dose (180-365 days, 366-540 days). Participants will be randomized in a 1:1 ratio to receive 1 dose of the ReCOV or placebo on Day 0.

SUMMARY:
Study Objective(s) To evaluate the safety, immunogenicity and protective efficacy of 1 dose of ReCOV in participants who have received 2 or 3 doses of inactivated SARS-CoV-2 vaccination in Chinese adults aged 18 years and older.

Primary objective To demonstrate the safety within 30 days after booster dose. Secondary objective(s) To evaluate the immunogenicity after booster dose. To demonstrate the safety within 6 months after booster dose. To evaluate the protective efficacy of RT-PCR-confirmed SARS-CoV-2 infection and COVID-19 after booster dose.

Indications：Prevention of COVID-19 caused by SARS-CoV-2 Population：Participants aged 18 years and older who completed 2 or 3 doses vaccination of inactivated COVID-19 vaccines and whose last dose was given 6-18 months, of which the elderly aged 60 years and older account for about 10% to 15%.

Sample Size：Approximately 3,300 participants

DETAILED DESCRIPTION:
Study Background Currently, the continued prevalence and mutation of SARS-CoV-2 variants has increased the urgency of optimizing the epidemic prevention strategy. Data from numerous studies show that booster vaccination with traditional COVID-19 vaccine can induce certain levels of antibodies and have a neutralizing effect on variants, which is the main means of responding to the current outbreak. By the end of November 2022, the booster vaccination rate of COVID-19 vaccine in China has exceeded 70%. However, recently, the surge in the number of infections and the strain on medical resources have made the task of the epidemic prevention increasingly difficult. The research and development of a new generation of COVID-19 vaccine with better broad-spectrum cross-neutralizing activity against endemic strains has become an important direction for the prevention of SARS-CoV-2 epidemics.

The recombinant two-component COVID-19 vaccine (CHO cell) developed and produced by Jiangsu Recbio Biotechnology Co., LTD. ( Recbio ), referred to as "ReCOV", is a new structurally designed COVID-19 vaccine guided by neutralizing antibodies. The antigen of ReCOV is selected from the amino acid sequence 14-541 (NTD and RBD structural domains) of Spike protein of SARS-CoV-2 prototype strain, and the foldon structural domain derived from T4 phage is fused at the C-terminus to form a trimerized protein containing NTD-RBD-foldon. For clinical use, a novel adjuvant BFA03 (similar to AS03 developed by GSK) consisting of squalene, α-tocopherol and polysorbate 80 is mixed to induce the body to produce specific neutralizing antibodies, block the binding of SARS-CoV-2 to the host, stimulate the body to produce anti-SARS-CoV-2 immunity, and is used to prevent the disease caused by SARS-CoV-2 infection. Non-clinical studies have shown that ReCOV was safe and well tolerated, with strong neutralizing effects against the prototype SARS-CoV-2 strain and multiple variants, and protection against SARS-CoV-2 attack.

To date, ReCOV's overseas clinical studies are actively underway. Among them, the phase I study of primary immunity has been completed, and three phase II studies of primary and sequential booster immunity will be completed in the near future for primary and interim analyses, respectively. The Phase III international multicenter study on the efficacy of primary immunity protection was initiated at the end of October 2022, and as of the preparation of this study protocol, more than 2,000 subjects have been enrolled and completed the first dose of vaccine, of which more than 1,000 have received two doses. During the same period, the ReCOV in-country Phase I study is ongoing. Phase I and II studies of ReCOV in both Caucasian and Asian populations showed good safety profiles, with no serious vaccine-related adverse events or adverse events leading to early study withdrawal reported, and the majority of adverse events were grade 1-2. Blinded data from the phase III study of primary immunization showed that the overall safety of ReCOV vaccination was good, and the safety characteristics were consistent with those of the phase I and II studies. The primary immunization study showed that two doses of ReCOV vaccination induced high levels of neutralizing antibodies against the prototype strain of the live virus and a significant Th1-biased cellular immune response with good immune persistence. Phase II studies of primary and sequential booster immunizations showed that ReCOV-induced neutralizing antibodies produced high levels of cross-neutralization against Omicron BA.2, BA.4/5, and BA.2.75 variants, with only 1.6 to 2.0-fold, 2.0 to 3.5-fold, and 2.6 to 3.0-fold decreases in titers compared to the prototype strain, respectively. Neutralizing antibody levels induced by the ReCOV sequential booster against the prototype strain and the Omicron BA.2, BA.4/5, and BA.2.75 variants were 10.8 to 17.3 times higher than the homologous booster of the control inactivated vaccine and significantly better than the heterologous booster immunization of the Pfizer mRNA vaccine.Data from all studies have shown that ReCOV is well tolerated and safe, with excellent immunogenicity and strong cross-protection against the current SARS-CoV-2 epidemic strain. Based on the previous clinical studies, this study will further evaluate the safety and immunogenicity of ReCOV booster immunization and explore its protective efficacy against SARS-CoV-2 infection and COVID-19 in Chinese population that has completed 2 or 3 doses of inactivated COVID-19 vaccine.

Study Design：This is a randomized, double-blind, placebo-controlled study to evaluate the safety, immunogenicity, and protective efficacy of a booster dose of ReCOV in a healthy Chinese population aged 18 years and older who have completed 2 or 3 doses of inactivated COVID-19 vaccine 6 to 18 months (180 to 540 days) after vaccination and who have been asked about their history of COVID-19 within the previous 6 months.Approximately 3300 participants will be enrolled, including an immunogenic subgroup of approximately 240. Approximately 10% to 15% of all subjects will be 60 years of age and older. Enrolled subjects will be stratified by age (18-59 years, 60 years and older), number of previous doses of COVID-19 vaccine (2 or 3 doses), and interval from the last previous dose (180-365 days, 366-540 days). Participants will be randomized in a 1:1 ratio to receive 1 dose of the ReCOV or placebo on Day 0.The study is divided into a screening period, a vaccination and follow-up period (randomization to 30 days after completion of booster immunization), and a long-term follow-up period (30 days after completion of booster immunization followed up to 6 months). At the end of the study vaccination and follow-up period, a first interim analysis (Interim Analysis, IA-1) of safety and available immunogenicity data will be performed. This will be followed by a 2nd interim analysis (Interim Analysis, IA-2) when at least 66.7% of the total number of target symptomatic COVID-19 endpoint cases have been collected (i.e., at least 103 symptomatic COVID-19 endpoint cases). Thereafter, a final analysis of safety, immunogenicity, and protective efficacy (Final Analysis, FA) will be performed after 6 months of follow-up after all subjects have completed booster immunization.

Safety observations All AEs within 30 minutes, solicited (local and systemic) AE within 7 days and unsolicited AE within 30 days after vaccination in all participants will be assessed. To assess the incidence, severity, and causality of SAEs and of AESI, and the occurrence of pregnancy events [newborns follow-up for at least 12 months after birth (female participant pregnancies and male participant partner pregnancies, mainly focus on newborn birth defects, abnormal growth and development, abnormal immune function and other events)], in all participants within 6 months after vaccination.

Solicited AE Solicited local AE：Pain、Pruritus、Redness、Swelling、Rash、Induration、Cellulitis Solicited systemic AE：Fatigue, fatigue, Fever, diarrhea, constipation, dysphagia, anorexia, vomiting, nausea, Myalgia(non-injection site), arthralgia, arthritis, headache, syncope, new seizures, cough, acute bronchospasm, dyspnea, pruritus at non vaccination sites (no skin damage), skin and mucous membrane abnormalities, insomnia, and acute allergic reaction.

Unsolicited AE All other AEs excluding Solicited AEs that occurred during the study. Immunogenicity observations For participants in immunogenicity subgroup, venous blood samples will be collected before the booster dose, 14 days, 3 months and 6 months after the booster dose vaccination.

Serum antibody (SARS-CoV-2 pseudo-virus neutralizing antibodies) titers of the SARS CoV-2 prototype strain and epidemic strain will be measured.

Protective efficacy observations From the time of the investigational vaccination, investigators are required to instruct subjects to use the SARS-CoV-2 antigen rapid test kit provided in this study and to perform 2 antigen tests per week for the first 3 months (2 tests should be separated by at least 2 days) and at least 1 antigen test per week thereafter (adjacent tests should be separated by at least 2 days), with the frequency of testing adjustable according to changes in the epidemic situation. The results of the antigen rapid test need to be photographed and sent to the investigator. Subjects with positive results are required to report immediately to the investigator, go to the nearest designated or approved SARS-CoV-2 nucleic acid sampling site on the same day under the direction of the investigator, collect two nasopharyngeal/oropharyngeal swabs at a time, and keep them in a sample tube for RT-PCR testing, and nucleic acid sequencing and genotyping in the central laboratory. When the RT-PCR test result is positive and the case is determined to be an endpoint case, the sample tube needs to be sent to the central laboratory for nucleic acid sequencing and genotype analysis. For subjects who tested positive for nucleic acid, the investigator is required to contact the subject for the next 3 days to collect and record the occurrence of the subject's COVID-19 symptoms. In addition, depending on the local epidemiological situation and epidemic prevention policies, investigators could instruct subjects to increase the frequency of antigen or nucleic acid testing.

Since the investigational vaccination, investigators are required to instruct subjects to promptly report symptoms that may be associated with COVID-19. If the subject reports any symptoms that may be associated with COVID-19, the investigator is instructed to promptly perform a SARS-CoV-2 antigen test or nucleic acid test. If the antigen or nucleic acid test is negative, investigators are required to instruct subjects to complete at least one subsequent antigen or nucleic acid test within 3 days, and subjects with a positive antigen test are required to complete nucleic acid sampling, testing and reporting of results, as well as sequencing and genotyping (if applicable) according to the process described above. The investigator may instruct subjects to increase the frequency of antigen or nucleic acid testing if necessary.

During the study, all subjects diagnosed with COVID-19 should be followed up by the investigator (at least twice a week) according to the study center's SOP for the management of COVID-19 positive cases until clinical outcome (i.e., asymptomatic for two consecutive days or death ) is achieved. If necessary, subjects should be evaluated for immunogenicity or additional testing, such as other inflammatory factors, target organ immunopathology, etc., to adequately assess for Antibody-Dependent Enhancement (ADE) or Vaccine Enhanced Disease (VED).

Study duration： Each subject takes approximately 6 months from enrollment to the final study visit .

Early exit criteria：1.The subject requests to withdraw from the study. 2.The subject has poor compliance and is unable to complete the follow-up in compliance with the protocol.

3.The subject is lost to follow-up and could not be reached after 3 or more attempts by the investigator to contact the subject.

4.Subjects is found to have violated the eligibility criteria during the study will be allowed to continue the study based on the investigator's judgment.

5.Other cases in which the investigator judges that it is not appropriate to continue participation in this study.

Study suspension or termination criteria Study suspension criteria If any participant vaccinated with the study vaccine (in any group) develops a Grade 4 AE or SAE after vaccination that is assessed as possibly related by the investigator.

≥15% of subjects developed a grade ≥3 AE possibly related to study vaccine that did not remit for 48 hours (note: "remission" is defined as an AE outcome of improvement, stable status, or return to severity below grade 3 with or without reasonable intervention by the investigator).

If one of the above suspension criteria occurs at any time during the study, the investigator is required to immediately suspend the trial and evaluate the appropriate safety event with the sponsor and the medical monitor. Subjects should not be given the study vaccine until the safety assessment has been completed. During this period, enrolled subjects will continue to be followed for safety, immunogenicity and protective efficacy as specified in the protocol.

Study termination criteria The sponsor makes a decision to terminate the trial early. AEs related to the study vaccine ≥ Grade 3 occurring in more than 30% of the participants.

In the occurrence of a grade ≥4 AE or SAE that may be related to the experimental vaccination, the investigator and sponsor will jointly discuss and decide whether to terminate the trial.

Termination at the request of IRB or administrative department In the event of early termination of the study, the sponsor will notify the investigator and the GCP immediately with the reasons as required by registration regulations.

Considering the possibility of changes in prevalence in the participating areas, the sample size estimates can be updated based on the prevalence in the participating areas prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

* 1.Adults aged 18 years and older. 2.Previous completion of 2 or 3 doses of inactivated COVID-19 vaccine and compliance with the vaccination procedures in the current instructions. The last dose of vaccination is 6 to 18 months (180 to 540 days, including the threshold) after the investigational vaccination, and proof of previous vaccination can be provided.

  3.Understand the content of the ICF, and voluntarily sign the ICF. 4.Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.

  5.Healthy participants or participants with mild underlying disease [in a stable state without exacerbation (no admission to hospital or no major adjustment to treatment regimen, etc.) for at least 3 months prior to enrollment in this study].

  6.Female participants
  * Surgically sterilized or ≥ 2 years post-menopause, or negative urine pregnancy test and willing to use effective contraception (e.g., condoms, IUDs) within 90 days of investigational vaccination. Contraceptive use is not allowed.
  * Consent to not breastfeed during the study and for at least 90 days after investigational vaccination。 male participants Subjects of childbearing potential who agree to use effective contraception (e.g., condoms, spermicide) within 90 days of study vaccination.

Exclusion Criteria:

* 1.Positive SARS-CoV-2 antigen during the screening period. 2.History of SARS, MERS, COVID-19 or known asymptomatic SARS-CoV-2 infection within 6 months prior to screening.

  3.Fever (axillary temperature ≥37.3 ℃) within 72 hours prior to vaccination. 4.History of severe allergy to any component of the experimental vaccine, including adjuvant components (squalene, alpha-tocopherol, and polysorbate 80, etc.), such as anaphylaxis, anaphylactic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, local anaphylactic necrotizing reaction (Arthus reaction); or previous history of severe side effects of any vaccine or drug, such as: allergy, urticaria, skin eczema, dyspnea, angioneurotic edema, etc.

  5.Currently suffering from acute infectious diseases or in the active stage of chronic infectious diseases, including but not limited to hepatitis B, hepatitis C.

  6.Current cancer, immune disorders (e.g., human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, absence of spleen or splenectomy, and other immune disorders that the investigator believes may have an impact on immune response), etc.; current other serious chronic diseases such as unstably controlled hypertension, asthma, heart disease, diabetes, liver or kidney disease, thyroid disease, hematologic system disorders (coagulation disorders or bleeding tendency), neurological/psychiatric disorders such as convulsions, epilepsy, etc.

  7.Undergoing anti-tuberculosis treatment. 8.Prolonged (defined as more than 14 days) use of immunosuppressive or other immunomodulatory drugs, anti-allergy therapy, or cytotoxic therapy within 6 months prior to the vaccine. Inhaled/nebulized, intra-articular, intradural, or topical (skin or eyes) corticosteroids are permitted. Topical doses should not exceed the recommended dose of the drug instructions.

  9.Have received blood products within 3 months prior to enrollment or plan to receive them during the study period.

  10.Participants who have received any other investigational product within 1 month prior to enrollment or intent to receive other investigational products during the study period.

  11.Received an inactivated vaccine or protein vaccine within 14 days prior to enrollment, or a live attenuated vaccine or adenovirus vector vaccine within 1 month, or intent to receive any other vaccine (except seasonal influenza vaccine or vaccine requiring emergency vaccination) during the study period.

Participants deemed unsuitable for participation in this study based on the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
solicited (local and systemic) AE | 7 days after booster dose
  Incidence of each solicited (local and systemic) AE within 7 days after booster dose.
unsolicited AE | within 30 days after booster dose
  Incidence of each unsolicited AE within 30 days after booster dose.
AE associated with investigational vaccine | within 30 days after booster dose
  Incidence of AE associated with investigational vaccine within 30 days after booster dose.

SECONDARY OUTCOMES:
Immunogenicity | on the 14th day, 3 months and 6 months after booster dose
  Immunogenicity：Geometric mean titer (GMT), Seroconversion Rate (SCR) and Geometric mean Increase (GMI) of neutralizing antibody responses against SARS CoV-2 prototype strain and epidemic strain on the 14th day, 3 months and 6 months after booster dose.
Safety observation | 6 months after booster dose
  Safety：Incidence of SAEs and AESIs from the day of booster dose to 6 months after booster dose.
protective efficacy | 14 days after booster dose
  protective efficacy：Number of RT-PCR confirmed, symptomatic COVID-19 cases (all severity levels) 14 days after booster dose.Number of RT-PCR-confirmed SARS-CoV-2 infection cases 14 days after booster dose.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No